CLINICAL TRIAL: NCT00955279
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Parallel-group, Placebo-controlled Study Evaluating the Safety and Efficacy of Treatment With Ustekinumab or Golimumab in Subjects With Chronic Sarcoidosis
Brief Title: A Study to Evaluate the Safety and Effectiveness of Ustekinumab or Golimumab Administered Subcutaneously (SC) in Patients With Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016405; 1275148SCD2001 (Other: Centocor); 2009-010714-30 (EudraCT Number)
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Sarcoidosis
Keywords: Ustekinumab; CNTO 1275; Stelara; Golimumab; CNTO 148; Simponi; Sarcoidosis; Sarcoid; Pulmonary Sarcoidosis; Skin Sarcoidosis
MeSH Terms: conditions — Sarcoidosis; Sarcoidosis, Pulmonary | interventions — golimumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Matching Placebo will be administered subcutaneously (injected under the skin by way of a needle) every 4 weeks up to Week 24.
  Interventions: Drug: Placebo
- Golimumab (Experimental): Golimumab will be administered subcutaneously at a dose of 200 milligram (mg) at Week 0 and thereafter at a dose of 100 mg every 4 weeks up to Week 24.
  Interventions: Drug: Golimumab
- Ustekinumab (Experimental): Ustekinumab will be administered subcutaneously at a dose of 180 mg at Week 0 and thereafter at a dose of 90 mg at Week 8, 16 and 24 and matching Placebo was administered subcutaneously at Week 4, 12 and 20.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Placebo — Matching Placebo will be administered subcutaneously (injected under the skin by way of a needle) every 4 weeks up to Week 24.
  Arms: Placebo
Drug: Golimumab — Golimumab will be administered subcutaneously at a dose of 200 milligram (mg) at Week 0 and thereafter at a dose of 100 mg every 4 weeks up to Week 24.
  Arms: Golimumab
Drug: Ustekinumab — Ustekinumab will be administered subcutaneously at a dose of 180 mg at Week 0 and thereafter at a dose of 90 mg at Week 8, 16 and 24 and matching Placebo was administered subcutaneously at Week 4, 12 and 20.
  Arms: Ustekinumab

SUMMARY:
This study tests the safety and effectiveness of ustekinumab or golimumab compared to placebo (placebo looks like the drugs being studied, but has no active ingredients). The purpose of this research study is to determine if ustekinumab or golimumab is safe and to determine its effects (good and bad) on patients with chronic sarcoidosis with pulmonary and/or skin involvement. Patients with pulmonary involvement constitute the primary population for analysis, and patients with skin involvement constitute the secondary population; a patient may be in both populations. The study will be conducted at approximately 40 sites globally.

DETAILED DESCRIPTION:
Ustekinumab is approved for dosing in patients with psoriasis and golimumab is approved for dosing in patients with rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. This study will use either drug in patients with chronic sarcoidosis. Ustekinumab and golimumab are being tested to see if they may be useful in treating chronic sarcoidosis. This study will compare the effects (both good and bad) of ustekinumab and golimumab to those of placebo. The purpose of this study is to evaluate the safety and effectiveness of ustekinumab and golimumab (administered as individual treatments) in patients with chronic sarcoidosis with lung and/or skin involvement who still have symptoms even though receiving current therapy. About 180 patients will take part in the study. While in this study, patients may not take part in any other medical research studies. Ustekinumab and golimumab are not approved by the national health authorities for treatment of chronic sarcoidosis; therefore, they can only be used in a research setting to treat this condition. The screening phase of the study, where the doctor will determine if a patient is eligible for the study, will last 1 to 4 weeks. Patients are put into 1 of 3 groups and each group will get a different treatment. The results of the golimumab group and the ustekinumab group are compared to placebo. Patients will either receive ustekinumab, golimumab or placebo. Placebo looks like ustekinumab and golimumab and is given in the same way, by injection, but contains no active drug. Patients will receive study agent until Week 24 and will continue to be followed through Week 44 for assessment of safety and any other effects after discontinuation of therapy. The patient will continue to take all sarcoidosis medication(s) at current, stable dose for the first part of the study. If the patient remained on a stable steroid dose from Week 0 through Week 16 of the study, the study doctor will begin to taper (lower) the steroid dose. The steroid taper will continue through to the end of the Week 28 visit. The patient will continue to take their other sarcoidosis medication(s) at the same dose for the rest of the study. An independent Data Monitoring Committee will be responsible for reviewing the safety data for the study. Patients will be in the study for about 48 weeks. The end of the study is defined as the last visit of the last patient. A site-specific substudy is being implemented to collect serum and lung samples from patients who are currently enrolled in this study. A separate protocol is being implemented to collect lung fluid and serum samples from normal, healthy subjects to be used as comparators for similar samples obtained in the 1275148SCD2001 substudy. Patients will be randomly assigned to 1 of 3 treatment groups: ustekinumab (180 mg at Week 0, followed by 90 mg at Weeks 8, 16, and 24 with placebo at Weeks 4, 12, and 20), golimumab (200 mg at Week 0, followed by 100 mg at Weeks 4, 8, 12, 16, 20, and 24) or placebo (at Weeks 0, 4, 8, 12, 16, 20, and 24) administered by SC injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have sarcoidosis with onset date of >=2 years prior to screening with at least 1 of the following: a. pulmonary sarcoidosis defined as 1) a diagnosis of sarcoidosis with evidence of lung parenchymal disease (Stage II, III or IV on chest radiograph), and 2) an FVC of >=45% and <=80% of predicted normal value at screening, and 3) an MRC dyspnea score of >2 at screening, and 4) a 6 minute walk distance between 100 to 550 meters at screening, and 5) <=15% absolute change in percent-predicted FVC at baseline relative to screening AND/OR b. skin sarcoidosis defined as 1) active chronic skin lesions for >=3 months either on face or elsewhere on body that have not resolved on current systemic and/or local therapy, and 2) have either: a single lesion of >=2 cm in longest dimension or multiple (3 or more) lesions with at least 1 lesion having a longest dimension of >=1 cm, and 3) have an SPGA score >=2 at screening
* have been receiving treatment with oral corticosteroids and/or 1 or more immunomodulators for >=3-month period immediately prior to screening
* on a stable dose of these medications for >=4 weeks before screening

Exclusion Criteria:

* Have a diagnosis of other significant respiratory disorder other than sarcoidosis that would complicate the evaluation of response to treatment
* Have a smoking history of >=20 pack years
* Have used an investigational drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer
* have received previous administration of a treatment with any other therapeutic agent targeted at reducing TNFalpha within 6 months or 5 half-lives of the agent, whichever is longer, prior to screening
* Patients who have previously received biologic anti-TNFalpha agents outside of the above period are allowed to enter the study
* Have previously used cyclophosphamide
* Have previously used or received local therapy (including local injections) within 3 months before the screening visit or used or received treatment with prescription topical creams within 1 month before the screening visit for treatment of sarcoidosis skin lesions
* Have used any therapeutic agent targeted at reducing IL-12 and/or IL-23, including but not limited to, ustekinumab and briakinumab within 6 months or 5 half-lives of the agent, whichever is longer, prior to the screening visit
* have received natalizumab or agents that deplete or modulate the activity of B cells or T cells within 12 months of screening, or, if after receiving these agents, evidence is available at screening of persistent depletion of the targeted lymphocyte population
* have used any antibody (monoclonal or polyclonal) or antibody-based agents <= 6 months or within 5 half-lives of the biologic prior to the screening visit, whichever is longer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (53):
- United States (24):
  - Birmingham, Alabama
  - Los Angeles, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Chicago, Illinois
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Spartanburg, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Colchester, Vermont
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Denmark (4):
  - Aarhus
  - Arhus C
  - Hellerup
  - København NV
- France (5):
  - Bobigny
  - Lille
  - Marseille
  - Montpellier
  - Paris
- Germany (6):
  - Bad Berka
  - Berlin
  - Essen
  - Freiburg im Breisgau
  - Hanover
  - München
- Netherlands (3):
  - Amsterdam-Zuidoost
  - Rotterdam
  - Sittard
- Norway (2):
  - Oslo
  - Trondheim
- Bucharest, Romania
- United Kingdom (5):
  - Bristol
  - London
  - Portsmouth
  - Sheffield
  - Southampton

REFERENCES:
- [Derived] Judson MA, Mack M, Beaumont JL, Watt R, Barnathan ES, Victorson DE. Validation and important differences for the Sarcoidosis Assessment Tool. A new patient-reported outcome measure. Am J Respir Crit Care Med. 2015 Apr 1;191(7):786-95. doi: 10.1164/rccm.201410-1785OC. PMID 25594886
- [Derived] Crommelin HA, Vorselaars AD, van Moorsel CH, Korenromp IH, Deneer VH, Grutters JC. Anti-TNF therapeutics for the treatment of sarcoidosis. Immunotherapy. 2014;6(10):1127-43. doi: 10.2217/imt.14.65. PMID 25428650
- [Derived] Judson MA, Baughman RP, Costabel U, Drent M, Gibson KF, Raghu G, Shigemitsu H, Barney JB, Culver DA, Hamzeh NY, Wijsenbeek MS, Albera C, Huizar I, Agarwal P, Brodmerkel C, Watt R, Barnathan ES. Safety and efficacy of ustekinumab or golimumab in patients with chronic sarcoidosis. Eur Respir J. 2014 Nov;44(5):1296-307. doi: 10.1183/09031936.00000914. Epub 2014 Jul 17. PMID 25034562

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching Placebo was administered subcutaneously (injected under the skin by way of a needle) every 4 weeks up to Week 24.
- Golimumab: Golimumab was administered subcutaneously at a dose of 200 milligram (mg) at Week 0 and thereafter at a dose of 100 mg every 4 weeks up to Week 24.
- Ustekinumab: Ustekinumab was administered subcutaneously at a dose of 180 mg at Week 0 and thereafter at a dose of 90 mg at Week 8, 16 and 24 and matching Placebo was administered subcutaneously at Week 4, 12 and 20.
Period: Overall Study
Arm/Group | Placebo | Golimumab | Ustekinumab
Started | 58 | 55 | 60
Completed | 55 | 51 | 52
Not Completed | 3 | 4 | 8
Not completed — Other | 0 | 0 | 3
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Golimumab | Ustekinumab | Total
Number analyzed (Participants) | 58 | 55 | 60 | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (9.51) | 50.0 (9.44) | 49.8 (10.17) | 49.8 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 29 | 85
  Male | 29 | 28 | 31 | 88
Number of Participants by stratification factors [Number; unit: participants] — Participant allocation to treatment group was performed by interactive voice response system (IVRS) using a permuted block randomization stratified by baseline disease organ involvement (participants with pulmonary involvement only, participants with skin involvement only, and participants with both pulmonary and skin involvement) and prior use of anti-Tumor necrosis factor (TNF) biological therapy (yes or no).
  participants
    Both Pulmonary and Skin | 6 | 4 | 7 | 17
    Pulmonary Only | 38 | 38 | 39 | 115
    Skin Only | 14 | 13 | 14 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent-predicted Forced Vital Capacity (FVC) at Week 16
Description: Forced vital capacity (FVC) is a standard pulmonary function test used to quantify respiratory muscle weakness . FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%. Change was calculated as the value at Week 16 minus the baseline value.
Time Frame: Baseline (Day 1) and Week 16
Population: Modified intent-to-treat (mITT) population included all the participants who were randomized and who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: percent of predicted FVC
Arm/Group | Placebo | Golimumab | Ustekinumab
Number analyzed (Participants) | 44 | 42 | 46
percent of predicted FVC | 2.02 (1.350) | 1.15 (1.413) | -0.15 (1.279)
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority or Other; p = 0.543, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab; Test type: Superiority or Other; p = 0.126, ANCOVA

2. Secondary Outcome: Change From Baseline in 6-minute Walk Distance at Week 28
Description: Change from Baseline in 6-minute walk distance at Week 28 was calculated as 6-minute walk distance at Week 28 minus 6-minute walk distance at Baseline. The 6-minute walk distance was the total distance walked during the 6-minute walk test.
Time Frame: Baseline (Day 1) and Week 28
Population: mITT population included all the participants who were randomized and who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Placebo | Golimumab | Ustekinumab
Number analyzed (Participants) | 44 | 42 | 46
meters | 14.52 (14.223) | 12.53 (14.919) | -13.22 (13.584)
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority or Other; p = 0.896, Linear Contrasts Test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab; Test type: Superiority or Other; p = 0.063, Linear Contrasts Test

3. Secondary Outcome: Change From Baseline in the St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 28
Description: St. George's Respiratory Questionnaire (SGRQ) is a health related quality of life questionnaire consisting of 51 items in three components: symptoms, activity, and impacts. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life. Change from Baseline was calculated as the value at Week 28 minus value at Baseline.
Time Frame: Baseline (Day 1) and Week 28
Population: mITT population included all the participants who were randomized and who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Golimumab | Ustekinumab
Number analyzed (Participants) | 44 | 42 | 46
Units on a scale | -9.50 (2.790) | -6.86 (2.921) | -4.25 (2.662)
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority or Other; p = 0.374, Linear Contrasts Test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab; Test type: Superiority or Other; p = 0.073, Linear Contrasts Test

4. Secondary Outcome: Percentage of Responders With a Score of Less Than or Equal to 1 on Skin Physician's Global Assessment (SPGA) Scale
Description: The SPGA is 7-point scale used to assess the condition of skin in participants. The physician checks the state of the skin and gives them score from 0 (clear) to 5 (severe). Higher scores indicate worsening of skin condition.
Time Frame: Week 28
Population: Secondary population included all the participants with chronic sarcoidosis with skin involvement who have received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Golimumab | Ustekinumab
Number analyzed (Participants) | 20 | 17 | 21
Percentage of Participants | 30.0 (2.790) | 52.9 (2.921) | 14.3 (2.662)
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority or Other; p = 0.1931, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab; Test type: Superiority or Other; p = 0.2772, Fisher Exact

5. Secondary Outcome: Change From Baseline in Percent-predicted Forced Vital Capacity (FVC) at Week 28
Description: Forced vital capacity (FVC) is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%. Change is calculated as the value at week 28 minus the baseline value.
Time Frame: Baseline (Day 1) and Week 28
Population: mITT population included all the participants who were randomized and who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: percent of predicted FVC
Arm/Group | Placebo | Golimumab | Ustekinumab
Number analyzed (Participants) | 44 | 42 | 46
percent of predicted FVC | 1.59 (1.621) | 0.29 (1.697) | 0.56 (1.536)
Statistical Analysis 1: Comparison: Placebo vs Golimumab; Test type: Superiority or Other; p = 0.451, Linear Contrast Test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab; Test type: Superiority or Other; p = 0.546, Linear Contrast Test

ADVERSE EVENTS:
Time Frame: Baseline and Week 16
Arm/Group | Placebo | Golimumab | Ustekinumab
Serious Adverse Events (participants affected / at risk) | 9/58 | 7/55 | 10/60
Other Adverse Events (participants affected / at risk) | 52/58 | 49/55 | 52/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=58) | Golimumab (N=55) | Ustekinumab (N=60)
Bronchitis (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Psychiatric evaluation (Investigations) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral sarcoidosis (Nervous system disorders) | 1 | 0 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=58) | Golimumab (N=55) | Ustekinumab (N=60)
Abdominal Pain (Gastrointestinal disorders) | 3 | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 6 | 9
Nausea (Gastrointestinal disorders) | 6 | 7 | 8
Vomiting (Gastrointestinal disorders) | 7 | 4 | 6
Chest Discomfort (General disorders) | 0 | 1 | 3
Chills (General disorders) | 0 | 1 | 3
Fatigue (General disorders) | 8 | 11 | 12
Influenza Like Illness (General disorders) | 3 | 2 | 3
Injection Site Erythema (General disorders) | 0 | 4 | 1
Injection Site Pain (General disorders) | 1 | 3 | 1
Injection Site Pruritus (General disorders) | 1 | 3 | 0
Malaise (General disorders) | 0 | 0 | 3
Non-Cardiac Chest Pain (General disorders) | 5 | 0 | 0
Oedema Peripheral (General disorders) | 5 | 8 | 4
Pyrexia (General disorders) | 3 | 4 | 5
Sarcoidosis (Immune system disorders) | 3 | 4 | 10
Bronchitis (Infections and infestations) | 8 | 7 | 8
Herpes Zoster (Infections and infestations) | 3 | 1 | 2
Influenza (Infections and infestations) | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 9
Oral Herpes (Infections and infestations) | 3 | 0 | 1
Respiratory Tract (Infections and infestations) | 2 | 4 | 3
Sinusitis (Infections and infestations) | 9 | 3 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 13 | 6 | 10
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 4
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 3
Weight Increased (Investigations) | 3 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 | 0 | 0
Gout (Metabolism and nutrition disorders) | 3 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 13 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 9
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 5
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 11 | 3 | 8
Burning Sensation (Nervous system disorders) | 0 | 1 | 3
Headache (Nervous system disorders) | 12 | 7 | 12
Migraine (Nervous system disorders) | 3 | 1 | 0
Depression (Psychiatric disorders) | 3 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 11 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 7
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 6 | 6
Skin Lesion (Skin and subcutaneous tissue disorders) | 8 | 1 | 6
Hypertension (Vascular disorders) | 3 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days